CLINICAL TRIAL: NCT03103087
Title: LIBERTY 2: An International Phase 3 Randomized, Double-Blind, Placebo-Controlled Efficacy and Safety Study to Evaluate Relugolix Co-Administered With and Without Low-Dose Estradiol and Norethindrone Acetate in Women With Heavy Menstrual Bleeding Associated With Uterine Fibroids
Brief Title: LIBERTY 2: Efficacy & Safety Study of Relugolix in Women With Heavy Menstrual Bleeding Associated With Uterine Fibroids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Myovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MVT-601-3002; 2016-005113-50 (EudraCT Number)
Record Dates: First submitted 2017-02-08; First posted 2017-04-06 (Actual); Results first posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2021-09

CONDITIONS: Heavy Menstrual Bleeding; Uterine Fibroid
Keywords: Uterine Fibroid; Heavy Menstrual Bleeding; Menstrual Blood Volume
MeSH Terms: conditions — Menorrhagia; Leiomyoma | interventions — relugolix; estradiol, norethindrone drug combination; Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Relugolix plus E2/NETA (Group A) (Experimental): Relugolix co-administered with E2/NETA for 24 weeks.
  Interventions: Drug: Relugolix; Drug: Estradiol/norethindrone acetate
- Relugolix plus Delayed E2/NETA (Group B) (Experimental): Relugolix co-administered with E2/NETA placebo for 12 weeks, followed by relugolix co-administered with E2/NETA for 12 weeks.
  Interventions: Drug: Relugolix; Drug: Estradiol/norethindrone acetate; Drug: Estradiol/norethindrone acetate placebo
- Placebo (Group C) (Placebo Comparator): Relugolix placebo co-administered with E2/NETA placebo for 24 weeks.
  Interventions: Drug: Relugolix placebo; Drug: Estradiol/norethindrone acetate placebo

INTERVENTIONS:
Drug: Relugolix — Relugolix (40 mg) tablet administered orally once daily.
  Other Names: TAK-385; MVT-601
  Arms: Relugolix plus Delayed E2/NETA (Group B); Relugolix plus E2/NETA (Group A)
Drug: Estradiol/norethindrone acetate — E2 (1.0 mg)/NETA (0.5 mg) co-formulated capsule administered orally once daily.
  Other Names: E2/NETA; low-dose hormonal add-back
  Arms: Relugolix plus Delayed E2/NETA (Group B); Relugolix plus E2/NETA (Group A)
Drug: Relugolix placebo — Relugolix (0 mg) placebo tablet administered orally once daily and manufactured to match the relugolix tablet in size, shape, color, and odor.
  Arms: Placebo (Group C)
Drug: Estradiol/norethindrone acetate placebo — E2 (0 mg)/NETA (0 mg) placebo capsule administered orally once daily and designed to match the capsule containing E2/NETA in size, shape, color, and odor.
  Other Names: E2/NETA placebo
  Arms: Placebo (Group C); Relugolix plus Delayed E2/NETA (Group B)

SUMMARY:
The purpose of this study is to determine the benefit of relugolix 40 milligrams (mg) once a day co-administered with estradiol (E2) 1 mg and norethindrone acetate (NETA) 0.5 mg compared with placebo for 24 weeks on heavy menstrual bleeding associated with uterine fibroids.

DETAILED DESCRIPTION:
This study is an international phase 3 randomized, double-blind, placebo-controlled efficacy and safety study to evaluate 24 weeks of oral daily relugolix 40 mg co-administered with low-dose E2 and NETA (Group A) and 12 weeks of daily oral relugolix 40 mg alone followed by 12 weeks of daily oral relugolix 40 mg co-administered with low-dose E2 and NETA (Group B) compared with 24 weeks of placebo (Group C).

All participants completing the Week 24 visit, including participants randomized to placebo, were offered the opportunity to enroll in an open-label extension study in which all eligible participants will receive relugolix co-administered with low-dose E2 and NETA. Participants who did not enroll into the extension study had a follow-up visit approximately 30 days after the end of treatment (that is, after the participant's last dose of study medication).

Safety will be assessed throughout the study by monitoring adverse events, vital signs, physical examinations, clinical laboratory tests, 12-lead electrocardiograms, and assessments of bone mineral density.

ELIGIBILITY:
Key Inclusion Criteria:

1. Premenopausal female aged 18 to 50 years old (inclusive) on the day of signing and dating the informed consent form.
2. Has regularly occurring menstrual periods of ≤ 14 days duration with a cycle of 21 to 38 days from the start of 1 menstrual period until the start of the next, by participant history for at least 3 months prior to the first screening visit.
3. Has a diagnosis of uterine fibroids that is confirmed by a transvaginal and/or transabdominal ultrasound performed during the screening period.
4. Has heavy menstrual bleeding associated with uterine fibroids as evidenced by an MBL of ≥ 160 milliliter (mL) during 1 cycle or ≥ 80 mL per cycle for 2 menstrual cycles as measured by the alkaline hematin method during the screening period.

Key Exclusion Criteria:

1. Has transvaginal and/or transabdominal ultrasound during the screening period demonstrating pathology other than uterine fibroids that could be responsible for or contributing to the participant's heavy menstrual bleeding.
2. Has known rapidly enlarging uterine fibroids in the opinion of the investigator.
3. Has a weight that exceeds the weight limit of the DXA scanner or has a condition that precludes an adequate DXA measurement at the lumbar spine and proximal femur.
4. Has a history of or currently has osteoporosis, or other metabolic bone disease, hyperparathyroidism, hyperprolactinemia, hyperthyroidism, anorexia nervosa, or low traumatic (from the standing position) or atraumatic fracture (toe, finger, skull, face and ankle fractures are allowed). A history of successfully treated hyperparathyroidism, hyperprolactinemia, or hyperthyroidism is allowed if the participant's bone mineral density is within normal limits.
5. Has a history of the use of bisphosphonates, calcitonin, calcitriol, ipriflavone, teriparatide, denosumab, or any medication other than calcium and vitamin D preparations to treat bone mineral density loss.
6. Has been a participant in an investigational drug or device study within the 1 month prior to the first screening visit.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 382 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2020-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myovant Medical Monitor, Study Director — Myovant Sciences
Locations (117):
- United States (82):
  - Birmingham, Birmingham, Alabama
  - Mesa, Mesa, Arizona
  - Tucson, Tucson, Arizona
  - Tuscon, Tucson, Arizona
  - Canoga Park, Canoga Park, California
  - Huntington Beach, Huntington Beach, California
  - Long Beach, Long Beach, California
  - Los Angeles, Los Angeles, California
  - Panorama, Panorama City, California
  - San Diego, San Diego, California
  - Upland, Upland, California
  - Denver, Denver, Colorado
  - Lakewood, Lakewood, Colorado
  - Washington, Washington D.C., District of Columbia
  - Aventura, Aventura, Florida
  - DeLand, DeLand, Florida
  - Ft. Lauderdale, Fort Lauderdale, Florida
  - Jupiter, Jupiter, Florida
  - Lake City, Lake City, Florida
  - Loxahachee, Loxahatchee Groves, Florida
  - Miami, Miami, Florida
  - Miami Springs, Miami Springs, Florida
  - New Port Richey, New Port Richey, Florida
  - North Miami, North Miami, Florida
  - Oviedo, Oviedo, Florida
  - Plantation, Plantation, Florida
  - Port St. Lucie, Port Saint Lucie, Florida
  - Saint Cloud, Saint Cloud, Florida
  - Sarasota, Sarasota, Florida
  - Stuart, Stuart, Florida
  - Tampa, Tampa, Florida
  - Wellington, Wellington, Florida
  - West Palm Beach, West Palm Beach, Florida
  - Atlanta, Atlanta, Georgia
  - Decatur, Decatur, Georgia
  - Duluth, Duluth, Georgia
  - Norcross, Norcross, Georgia
  - Sandy Springs, Sandy Springs, Georgia
  - Savannah, Savannah, Georgia
  - Idaho Falls, Idaho Falls, Idaho
  - Nampa, Nampa, Idaho
  - Champaign, Champaign, Illinois
  - Chicago, Chicago, Illinois
  - Naperville, Naperville, Illinois
  - Oakbrook, Oak Brook, Illinois
  - Avon, Avon, Indiana
  - Shawnee, Shawnee Mission, Kansas
  - Marrero, Marrero, Louisiana
  - Metairie, Metairie, Louisiana
  - New Orleans, New Orleans, Louisiana
  - Baltimore, Baltimore, Maryland
  - Towson, Towson, Maryland
  - Bay City, Bay City, Michigan
  - Canton, Canton, Michigan
  - Detroit, Detroit, Michigan
  - Saginaw, Saginaw, Michigan
  - Norfolk, Norfolk, Nebraska
  - Las Vegas, Las Vegas, Nevada
  - New Brunswick, New Brunswick, New Jersey
  - Albuquerque, Albuquerque, New Mexico
  - Brooklyn, Brooklyn, New York
  - New York, New York, New York
  - Rochester, Rochester, New York
  - Durham, Durham, North Carolina
  - Raleigh, Raleigh, North Carolina
  - Winston Salem, Winston-Salem, North Carolina
  - Cincinnati, Cincinnati, Ohio
  - Columbus, Columbus, Ohio
  - West Reading, West Reading, Pennsylvania
  - Charleston, Charleston, South Carolina
  - Beaumont, Beaumont, Texas
  - Dallas, Dallas, Texas
  - Fort Worth, Fort Worth, Texas
  - Frisco, Frisco, Texas
  - Houston, Houston, Texas
  - Longview, Longview, Texas
  - San Antonio, San Antonio, Texas
  - Virginia Beach, Norfolk, Virginia
  - Richmond, Richmond, Virginia
  - Covington, Covington, Washington
  - Puyallup, Puyallup, Washington
  - Spokane, Spokane, Washington
- Belgium (4):
  - Brussels, Brussels
  - Ghent, Ghent
  - Jette, Jette
  - La Louvière, La Louvière
- Brazil (3):
  - Botucatu, Botucatu
  - Porto Alegre, Porto Alegre
  - São Paulo, São Paulo
- Chile (3):
  - Santiago, Santiago, Providencia
  - San Ramon, San Ramón
  - Santiago, Santiago
- Czechia (6):
  - Ceské Budejovice, České Budějovice
  - Jihlava, Jihlava
  - Nachod, Náchod
  - Olomouc, Olomouc
  - Ostrava, Ostrava
  - Pisek, Písek
- Hungary (8):
  - Debrecen, Debrecen, Hajdu
  - Nyíregyháza, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Budapest, Budapest
  - Debrecen, Debrecen
  - Gyula, Gyula
  - Kecskemét, Kecskemét
  - Pecs, Pécs
  - Szentes, Szentes
- Poland (7):
  - Poznan, Poznan, Greater Poland Voivodeship
  - Krakow, Krakow, Lesser Poland Voivodeship
  - Rzeszów, Rzeszów, Masovian Voivodeship
  - Białystok, Bialystok, Podlaskie Voivodeship
  - Bialystok, Bialystok, Podlaskie Voivodeship
  - Katowice, Katowice, Silesian Voivodeship
  - Gdańsk, Gdansk
- South Africa (4):
  - Cape Town, Cape Town, Western Cape
  - Bloemfontein, Bloemfontein
  - Centurion, Centurion
  - Parow, Parow

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Catherino WH, Al-Hendy A, Zaim S, Bouzegaou N, Venturella R, Stewart EA, Wu R, Vannuccini S, Perry JS, Rakov VG, Munro MG. Efficacy and safety of relugolix combination therapy in women with uterine fibroids and adenomyosis: subgroup analysis of LIBERTY 1 and LIBERTY 2. Fertil Steril. 2025 Sep;124(3):523-533. doi: 10.1016/j.fertnstert.2025.04.037. Epub 2025 May 2. PMID 40320117
- [Derived] Stewart EA, Lukes AS, Venturella R, Ferreira JA, Li Y, Hunsche E, Wagman RB, Al-Hendy A. A plain language summary describing changes in pain associated with uterine fibroids among women receiving relugolix combination therapy. Pain Manag. 2024 Sep;14(9):469-476. doi: 10.1080/17581869.2024.2408114. Epub 2024 Oct 28. PMID 39466126
- [Derived] Stewart EA, Al-Hendy A, Lukes AS, Madueke-Laveaux OS, Zhu E, Proehl S, Schulmann T, Marsh EE. Relugolix combination therapy in Black/African American women with symptomatic uterine fibroids: LIBERTY Long-Term Extension study. Am J Obstet Gynecol. 2024 Feb;230(2):237.e1-237.e11. doi: 10.1016/j.ajog.2023.10.030. Epub 2023 Oct 18. PMID 37863160
- [Derived] Al-Hendy A, Lukes AS, Venturella R, Villarroel C, McKain L, Li Y, Wagman RB, Stewart EA. A plain language summary of the long-term relugolix combination therapy study for uterine fibroids. J Comp Eff Res. 2023 Aug;12(8):e230069. doi: 10.57264/cer-2023-0069. Epub 2023 Jul 21. PMID 37477173
- [Derived] Al-Hendy A, Lukes AS, Poindexter AN 3rd, Venturella R, Villarroel C, Critchley HO, Li Y, McKain L, Arjona Ferreira JC, Langenberg AG, Wagman RB, Stewart EA. A plain language summary of the safety of relugolix combination therapy and improvement in symptoms in women with uterine fibroids from the LIBERTY 1 and LIBERTY 2 studies. Pain Manag. 2023 Apr;13(4):205-211. doi: 10.2217/pmt-2022-0085. Epub 2023 May 15. PMID 37183454
- [Derived] Al-Hendy A, Lukes AS, Poindexter AN 3rd, Venturella R, Villarroel C, McKain L, Li Y, Wagman RB, Stewart EA. Long-term Relugolix Combination Therapy for Symptomatic Uterine Leiomyomas. Obstet Gynecol. 2022 Dec 1;140(6):920-930. doi: 10.1097/AOG.0000000000004988. Epub 2022 Nov 2. PMID 36357960
- [Derived] Stewart EA, Lukes AS, Venturella R, Arjona Ferreira JC, Li Y, Hunsche E, Wagman RB, Al-Hendy A. Relugolix Combination Therapy for Uterine Leiomyoma-Associated Pain in the LIBERTY Randomized Trials. Obstet Gynecol. 2022 Jun 1;139(6):1070-1081. doi: 10.1097/AOG.0000000000004787. Epub 2022 May 2. PMID 35675604
- [Derived] Hunsche E, Rakov V, Scippa K, Witherspoon B, McKain L. The Burden of Uterine Fibroids from the Perspective of US Women Participating in Open-Ended Interviews. Womens Health Rep (New Rochelle). 2022 Mar 4;3(1):286-296. doi: 10.1089/whr.2021.0086. eCollection 2022. PMID 35415708
- [Derived] Al-Hendy A, Lukes AS, Poindexter AN 3rd, Venturella R, Villarroel C, Critchley HOD, Li Y, McKain L, Arjona Ferreira JC, Langenberg AGM, Wagman RB, Stewart EA. Treatment of Uterine Fibroid Symptoms with Relugolix Combination Therapy. N Engl J Med. 2021 Feb 18;384(7):630-642. doi: 10.1056/NEJMoa2008283. PMID 33596357

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 99 study centers throughout the world, including centers in the United States, Belgium, Brazil, Chile, Czech Republic, Hungary, Poland, and South Africa.
Pre-assignment Details: A total of 382 premenopausal women aged 18 to 50 years old (inclusive) with heavy menstrual bleeding (≥ 160 milliliters [mL] during 1 cycle or ≥ 80 mL per cycle for 2 menstrual cycles as measured by the alkaline hematin method) associated with uterine fibroids were randomized. One participant was randomized in error before eligibility confirmed.
Groups:
- Relugolix Plus Estradiol (E2])/Norethindrone Acetate (NETA) (Group A): Relugolix 40 milligrams (mg) co-administered with E2 (1.0 mg) and NETA (0.5 mg) for 24 weeks.
- Relugolix Plus Delayed E2/NETA (Group B): Relugolix 40 mg co-administered with placebo for E2/NETA for 12 weeks followed by relugolix 40 mg co-administered with E2/NETA (1.0/0.5 mg) for 12 weeks.
- Placebo (Group C): Placebo for relugolix co-administered with placebo for E2/NETA for 24 weeks.
Period: Overall Study
Arm/Group | Relugolix Plus Estradiol (E2])/Norethindrone Acetate (NETA) (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Started | 126 | 127 | 129
Completed | 102 | 98 | 102
Not Completed | 24 | 29 | 27
Not completed — Did not receive any study drug | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 1
Not completed — Lack of Efficacy | 2 | 1 | 1
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Adverse Event | 2 | 15 | 6
Not completed — Withdrawal by Subject | 13 | 6 | 6
Not completed — Lost to Follow-up | 4 | 2 | 7
Not completed — Other reason not reported | 1 | 3 | 5

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled and randomized in the study.
Groups:
- Relugolix Plus E2/NETA (Group A): Relugolix 40 mg co-administered with E2 (1.0 mg) and NETA (0.5 mg) for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C) | Total
Number analyzed (Participants) | 126 | 127 | 129 | 382
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 126 | 127 | 129 | 382
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (5.37) | 42.1 (5.25) | 41.8 (5.26) | 42.1 (5.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 127 | 129 | 382
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 34 | 32 | 84
  Not Hispanic or Latino | 106 | 91 | 96 | 293
  Unknown or Not Reported | 2 | 2 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 1 | 3
  Asian | 0 | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 63 | 66 | 74 | 203
  White | 58 | 50 | 49 | 157
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 4 | 5 | 4 | 13
Region of Enrollment [Number; unit: participants]
  Hungary | 7 | 7 | 8 | 22
  Belgium | 0 | 3 | 1 | 4
  United States | 94 | 94 | 96 | 284
  Czechia | 4 | 2 | 3 | 9
  Poland | 7 | 6 | 4 | 17
  Brazil | 1 | 3 | 1 | 5
  South Africa | 7 | 3 | 7 | 17
  Chile | 6 | 9 | 9 | 24
Mean MBL Volume [Mean (Standard Deviation); unit: mL] | 247.62 (185.553) | 227.41 (34.350) | 211.75 (129.903) | 228.45 (152.205)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Of Participants Who Achieved A Menstrual Blood Loss (MBL) Volume Of < 80 mL And A ≥ 50% Reduction From Baseline MBL Volume With Relugolix Plus E2/NETA
Description: A responder was a participant who had MBL volume of < 80 mL and at least a 50% reduction from baseline MBL volume over the last 35 days of treatment (up to Week 24). All returned feminine products collected at each clinical visit were analyzed by the alkaline hematin method to obtain the MBL volume. MBL volume was measured over the Week 24/early termination feminine product collection interval (up to 35 days prior to the last dose of treatment). The percentage of participants who were responders are presented.
  As per the objective of the study, the pre-specified primary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms are presented.
Time Frame: From Baseline up to the last 35 days of treatment (up to Week 24)
Population: All randomized participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 125 | 129
Percentage of participants | 71.2 [62.42 to 78.95] | 14.73 [9.11 to 22.04]
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was stratified by baseline MBL volume (< 225 mL or ≥ 225 mL) and geographic region (North America or Rest of World). Assessed at a 2-sided α = 0.05 significance level; Treatment Difference = 56.47, 95% CI 2-sided [46.45 to 66.49] — Treatment difference is relugolix plus E2/NETA minus placebo

2. Secondary Outcome: Percentage Of Participants With Amenorrhea Over The Last 35 Days Of Treatment
Description: Amenorrhea was defined as meeting 1 of the following criteria for 2 consecutive visits:
  * No feminine product returned due to reported amenorrhea;
  * No feminine product returned due to reports of spotting/negligible bleeding coupled with electronic diary (e-Diary) data indicating infrequent non-cyclic bleeding/spotting;
  * Feminine product collection with a negligible observed MBL volume coupled with e-Diary data indicating infrequent non-cyclic bleeding/spotting.
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms are presented.
Time Frame: From Baseline up to last 35 days of treatment (up to Week 24)
Population: All randomized participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 125 | 129
Percentage of participants | 50.40 [41.32 to 59.46] | 3.10 [0.85 to 7.75]
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was based on Cochran-Mantel-Haenszel test stratified by Baseline MBL volume (< 225 mL, ≥ 225 mL) and geographic region (North America or Rest of World). Assessed at a 2-sided α = 0.05 significance level; Treatment difference was relugolix plus E2/NETA minus placebo. 95% confidence interval (CI) for the difference is based on the normal approximation; Treatment Difference = 47.3, 95% CI 2-sided [38.04 to 56.56]

3. Secondary Outcome: Percent Change From Baseline At Week 24 In MBL Volume
Description: MBL volume was measured using the alkaline hematin method. Least square (LS) means for test of difference is Relugolix plus E2/NETA minus Placebo based on mixed-effect model with treatment, visit, region, Baseline MBL, and treatment by visit interaction included as fixed effects.
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms are presented.
Time Frame: Baseline, Week 24
Population: All randomized participants who received any amount of study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 125 | 129
percent change | -84.3 [-95.0 to -73.6] | -15.1 [-25.8 to -4.3]
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p < 0.0001, Mixed Models Analysis — Treatment, visit, region, Baseline MBL and treatment by visit interaction included as fixed effects. Assessed at a 2-sided α = 0.05 significance; Treatment Difference = -69.2, 95% CI 2-sided [-84.1 to -54.3], Standard Error of Mean 7.58 — Treatment difference was relugolix plus E2/NETA minus placebo

4. Secondary Outcome: Percentage Of Participants With A Hemoglobin Level ≤ 10.5 g/dL At Baseline Who Achieved An Increase Of > 2 g/dL From Baseline At Week 24
Description: Blood samples were collected from participants for hemoglobin measurements. Percentages are based on number of participants with hemoglobin ≤ 10.5 gram (g)/deciliter (dL) at Baseline and reported at Week 24.
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA with placebo arms are presented.
Time Frame: From Baseline up to Week 24
Population: All randomized participants who received any amount of study drug and had analyzable study data at the specified timepoint.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 31 | 37
Percentage of participants | 61.29 [42.19 to 78.15] | 5.41 [0.66 to 18.19]
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value is based on Cochran-Mantel-Haenszel test stratified by Baseline MBL volume (< 225 mL, ≥ 225 mL). Assessed at a 2-sided α = 0.05 significance level; Treatment Difference = 55.88, 95% CI 2-sided [37.25 to 74.52] — Treatment difference is relugolix plus E2/NETA minus placebo. 95% CI for difference is based on the normal approximation

5. Secondary Outcome: Percentage Of Participants With A Maximum Numerical Rating Scale (NRS) Score ≤ 1 For Uterine Fibroid-Associated Pain Over The Last 35 Days Of Treatment
Description: Uterine fibroid-associated pain was assessed by a pain numerical rating scale (NRS). The pain NRS is a validated, single-item, self-reported measure, which asks respondents to rank their pain on an 11-point scale as follows: 0 (no pain), 1 to 3 (mild pain), 4 to 6 (moderate pain), and 7 to 10 (severe pain).
  Participants were asked to document, in an e-Diary, the worst pain associated with their uterine fibroids that they experienced during the last 24 hours, every day until the end of study drug administration. Pain evaluable participants, defined as those who had maximum NRS score ≥ 4 at baseline and had at least 28 days (80% of the last 35 days of treatment) of pain scores recorded in the e-Diary, were analyzed.
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms are presented.
Time Frame: From Baseline up to Week 24
Population: All randomized participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 68 | 82
percentage of participants | 47.06 [34.83 to 59.55] | 17.07 [9.66 to 26.98]
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Treatment Difference = 29.99, 95% CI 2-sided [15.6 to 44.38] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Percent Change From Baseline At Week 24 In Primary Uterine Fibroid Volume
Description: The volume of the primary uterine fibroid was measured by transvaginal or transabdominal ultrasound.
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms are presented.
Time Frame: Baseline Week 24
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 95 | 98
percent change | -17.4 [-29.1 to -5.7] | -7.4 [-19.1 to 4.2]
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p = 0.2153, ANCOVA — LS Means based on analysis of covariance model including treatment, randomization stratification factors, Baseline MBL volume (< 225 mL, ≥ 225 mL) and geographic region (North America, Rest of World), and Baseline values as covariate; Treatment Difference = -10, 95% CI 2-sided [-25.8 to 5.8], Standard Error of Mean 8.03

7. Secondary Outcome: Percent Change From Baseline At Week 24 In Uterine Volume
Description: The volume of the uterus was measured by transvaginal or transabdominal ultrasound.
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms are presented.
Time Frame: From Baseline up to Week 24
Population: All participants who were randomized to treatment and who received at least 1 dose of study drug and had evaluable data at the specified timepoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 95 | 100
percent change | -13.8 [-20.4 to -7.1] | -1.5 [-8.2 to 5.1]
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p = 0.0078, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Treatment Difference = -12.2, 95% CI 2-sided [-21.3 to -3.2], Standard Error of Mean 4.57

8. Secondary Outcome: Change From Baseline At Week 24 In UFS-QoL Bleeding And Pelvic Discomfort Scale Score As Measured By The UFS-QoL (Q1, Q2, Q5)
Description: The Uterine Fibroid Symptom and Health-Related Quality of Life (UFS-QoL) Bleeding and Pelvic Discomfort (BPD) Scale has been derived from the UFS-QoL Symptoms Scale. The scale consists of the following 3 symptoms proximal to uterine fibroids: Heavy bleeding during your menstrual period (Question [Q] 1), passing blood clots during your menstrual period (Q2), and feeling tightness or pressure in your pelvic area (Q5), raw scores were transformed to a normalized score: Transformed Score = [(Actual raw score - lowest possible raw score)/(Possible raw score range)]*100 Transformed score ranges from 0 to 100 based on Likert scale (None of time, a little of time, some of the time, most of the time and all of the time). Lower score indicates minimal symptom severity and higher score indicates symptom severity.
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms
Time Frame: Baseline Week 24
Population: All randomized participants who received any amount of study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 96 | 95
units on a scale | -51.7 [-57.4 to -46.0] | -18.3 [-24.1 to -12.6]
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p < 0.0001, Mixed Models Analysis — Assessed at a 2-sided α = 0.05 significance level; Treatment Difference = -33.4, 95% CI 2-sided [-41.2 to -25.5], Standard Error of Mean 3.98 — Relugolix plus E2/NETA minus placebo. Treatment, visit, region, Baseline MBL and treatment by visit interaction as fixed effects

9. Secondary Outcome: Percent Change From Baseline At Week 12 In Bone Mineral Density At The Lumbar Spine (L1 to L4) As Assessed By DXA
Description: Bone mineral density (BMD) was assessed by dual-energy x-ray absorptiometry (DXA) at the lumbar spine (L1, L2, L3, and L4) at Baseline and at Week 12. The scans were read by the central radiology laboratory in accordance with the imaging charter. The same DXA machine was used at the local imaging center at each site and operated in the same scan mode for all images procured for an individual participant. All images were submitted for central reading. The central radiology laboratory collected and evaluated all DXA scans for acceptability and measured BMD. The LS means were based on a mixed-effect model with visit, region, Baseline MBL volume, age at Baseline, body mass index at Baseline, BMD at Baseline, race, and treatment by visit interaction included as fixed effects.
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms are presented.
Time Frame: From Baseline up to Week 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B)
Number analyzed (Participants) | 103 | 95
percent change | -0.819 (0.2686) | -1.919 (0.2767)

10. Secondary Outcome: Percent Change From Baseline At Week 24 In Bone Mineral Density At The Lumbar Spine (L1 To L4), Total Hip, And Femoral Neck As Assessed By DXA
Description: BMD was assessed by DXA at the lumbar spine (L1, L2, L3, and L4), total hip, and femoral neck (same leg across participants) at Baseline and at Week 24. The scans were read by the central radiology laboratory in accordance with the imaging charter. The same DXA machine was used at the local imaging center at each site and operated in the same scan mode for all images procured for an individual participant. All images were submitted for central reading. The central radiology laboratory collected and evaluated all DXA scans for acceptability and measured BMD. The LS means were based on a mixed-effect model with visit, region, Baseline MBL volume, age at Baseline, body mass index at Baseline, BMD at Baseline, race, and treatment by visit interaction included as fixed effects. For Relugolix plus E2/NETA Lumbar Spine (L1 to L4), number (n)=95.
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only rel
Time Frame: Baseline through Week 24
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 98 | 95
percent change
  Lumbar Spine (L1-L4) | -0.126 (0.2971) | 0.315 (0.2909)
  Total Hip | -0.173 (0.2221) | -0.044 (0.2200)
  Femoral Neck | -0.684 (0.3730) | 0.019 (0.3697)

11. Secondary Outcome: Percentage Of Participants Experiencing Vasomotor Symptoms Through Week 12
Description: An adverse event was defined as an unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product, whether or not related to the medicinal product. The preferred terms of hyperhidrosis, feeling hot, hot flush, night sweats, and flushing were combined to describe vasomotor symptoms. Participants with multiple events for a given preferred term were counted only once for each preferred term. Reported confidence interval (CI) based on exact binomial 95% CI (Clopper-Pearson). As per the objective of the study, the secondary analysis compared relugolix plus E2/NETA with relugolix plus delayed E2/NETA at Week 12 and are presented below.
Time Frame: Baseline through Week 12
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B)
Number analyzed (Participants) | 126 | 126
percentage of participants | 5.56 [2.26 to 11.11] | 35.71 [27.38 to 44.74]
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Relugolix Plus Delayed E2/NETA (Group B); Test type: Other; p < 0.0001, Fisher Exact; Risk Ratio (RR) = 0.16, 95% CI 2-sided [0.07 to 0.33]

12. Secondary Outcome: Percentage Of Participants Experiencing Vasomotor Symptoms Through Week 24
Description: An adverse event was defined as an unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product, whether or not related to the medicinal product. The preferred terms of hyperhidrosis, feeling hot, hot flush, night sweats, and flushing were combined to describe vasomotor symptoms. Participants with multiple events for a given preferred term were counted only once for each preferred term.
  Reported percentages based on the total number of participants in each treatment group.
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms are presented.
Time Frame: Baseline through Week 24
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 126 | 129
percentage of participants | 6.3 | 3.9

13. Secondary Outcome: Predose Trough Concentrations Of Relugolix And NET In The Relugolix Plus E2/NETA Group At Week 24
Description: Blood samples for determination of relugolix and NET plasma concentrations were collected predose at Week 24. Relugolix and NET plasma concentrations were determined using validated bioanalytical methodology.
  Concentrations below the quantification limit (BQL) were set to 0 for analysis of summary statistics. As per the objective of the study, only relugolix plus E2/NETA concentration is presented.
Time Frame: Week 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Relugolix Plus E2/NETA (Group A)
Number analyzed (Participants) | 93
ng/mL
  Relugolix | 1.96 (2.025)
  NET | 0.28 (0.285)

14. Secondary Outcome: Predose Trough Concentrations Of E2 In The Relugolix Plus E2/NETA Group At Week 24
Description: as for outcome 13
Time Frame: Week 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Relugolix Plus E2/NETA (Group A)
Number analyzed (Participants) | 88
pg/mL | 45.34 (46.330)

15. Secondary Outcome: Change From Baseline At Week 24 In Predose Concentrations Of E2 In The Relugolix Plus E2/NETA Group
Description: Blood samples for determination of E2 serum concentrations were collected predose at Week 24. Relugolix and NET plasma concentrations were determined using validated bioanalytical methodology.
  Concentrations below the quantification limit (BQL) were set to 0 for analysis of summary statistics. As per the objective of the study, only relugolix plus E2/NETA concentration is presented.
Time Frame: Baseline, Week 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Relugolix Plus E2/NETA (Group A)
Number analyzed (Participants) | 93
pg/mL | -22.30 (66.552)

16. Secondary Outcome: Time To MBL Response
Description: Defined as the time to achieve an MBL volume of < 80 mL and a ≥ 50% reduction from Baseline MBL volume as measured by the alkaline hematin method.
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms are presented.
Time Frame: From Baseline through Week 24
Population: All participants who were randomized to treatment and who received at least 1 dose of study drug.
Measure: Median (97.5% Confidence Interval); unit: weeks
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 104 | 34
weeks | 8.4 [8.1 to 9.0] | 27.1 [25.0 to 27.4]
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p < 0.0001, Log Rank — P-value is based on Log-rank test stratified by Baseline MBL volume (< 225 mL, ≥ 225 mL) and geographic region (North America, Rest of World) from the proportional hazard regression model comparing relugolix plus E2/NETA with placebo

17. Secondary Outcome: Sustained Amenorrhea Rate (No Or Negligible Bleeding)
Description: Sustained amenorrhea is defined as participants time to achieve and maintain amenorrhea until the date of last study drug.
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms are presented.
Time Frame: Week 24
Population: All participants who were randomized to treatment and who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 125 | 129
Participants | 63 | 4
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value for testing difference between relugolix plus E2/NETA and placebo is based on Cochran-Mantel-Haenszel test stratified by Baseline MBL volume (< 225 mL, ≥ 225 mL) and geographic region (North America, Rest of World)

18. Secondary Outcome: Time To Achieving Sustained Amenorrhea (No Or Negligible Bleeding)
Description: Sustained amenorrhea status as determined based on time to achieve and maintain amenorrhea status.
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms are presented.
Time Frame: From Baseline through Week 24
Population: All participants who were randomized to treatment and who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 63 | 4
weeks | 16.3 [8.1 to NA] — Not evaluable. | NA [NA to NA] — Sustained amenorrhea was not reached.
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 16, analysis 1]

19. Secondary Outcome: Time To Achieving Amenorrhea (No Or Negligible Bleeding)
Description: Time to amenorrhea was defined as the weeks from date of first dose of study drug to the start of amenorrhea.
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms are presented.
Time Frame: From Baseline through Week 24
Population: All participants who were randomized to treatment and who received at least 1 dose of study drug and had analyzable data at the specified timepoint.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 71 | 11
weeks | 8.9 [5.3 to 16.3] | NA [NA to NA] — Amenorrhea was not reached.
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 16, analysis 1]

20. Secondary Outcome: Number Of Participants With Hemoglobin ≤ 10.5 g/dL At Baseline And Achieved An Increase Of > 2 g/dL At Week 24
Description: As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms are presented.
Time Frame: From Baseline through Week 24
Population: All participants who were randomized to treatment, received at least 1 dose of study drug, and had hemoglobin ≤ 10.5 g/dL at Baseline and an assessment at Week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 31 | 37
Participants | 19 | 2
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was based on Cochran-Mantel-Haenszel test stratified by Baseline MBL volume (< 225 mL, ≥ 225 mL)

21. Secondary Outcome: Percent Change From Baseline At Week 24 In Hemoglobin For Women With A Hemoglobin Concentration ≤ 10.5 g/dL At Baseline
Description: as for outcome 20
Time Frame: Baseline, Week 24
Population: All randomized participants who received any amount of study drug and had analyzable data at the specified timeframe.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 31 | 37
percent change | 24.3 (3.02) | 4.3 (2.68)
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p < 0.0001, Mixed Models Analysis — LS means and p-value for test of difference is relugolix plus E2/NETA minus Placebo based on mixed-effect model with treatment, visit, region, Baseline MBL and treatment by visit interaction included as fixed effects

22. Secondary Outcome: Number Of Participants With Hemoglobin Increase Of ≥ 1 g/dL From Baseline To Week 24 Among Those With Below Lower Limit Of Normal
Description: as for outcome 20
Time Frame: Week 24
Population: All randomized participants who received any amount of study drug and had analyzable data at the specified timeframe.
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 69 | 75
Participants | 35 | 18
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was based on Cochran-Mantel-Haenszel test stratified by Baseline MBL volume (< 225 mL, ≥ 225 mL) and geographic region (North America, Rest of World). Lower limit of normal is Hgb < 11.6 g/dL

23. Secondary Outcome: Change From Baseline At Week 24 In The UFS-QoL Symptom Severity Scale Score
Description: Transformed score ranges from 0 to 100 based on Likert scale (None of time, a little of time, some of time, most of the time and all of the time.) Lower score indicates minimal symptom severity and higher score indicates maximum symptom severity. A negative change from baseline indicates improvement.
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms are presented.
Time Frame: Baseline, Week 24
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 96 | 95
score on a scale | -36.1 (2.59) | -13.7 (2.61)
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p < 0.0001, Mixed Models Analysis — LS means and p-value for test of difference is relugolix plus E2/NETA minus placebo based on mixed-effect model with treatment, visit, region, Baseline MBL, and treatment by visit interaction included

24. Secondary Outcome: Change From Baseline At Week 24 In The UFS-QoL Activities Scale Score
Description: Transformed score ranges from 0 to 100 based on Likert scale (None of time, a little of time, some of the time, most of the time and all of the time). Higher scores are indicative of better health-related quality of life (high score = good).
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms are presented.
Time Frame: Baseline, Week 24
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 96 | 95
score on a scale | 43.6 (2.77) | 17.1 (2.80)
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p < 0.0001, Mixed Models Analysis — LS means and p-value for test of difference is relugolix plus E2/NETA minus placebo based on mixed-effect model with treatment, visit, region, Baseline MBL, and treatment by visit interaction included as fixed effects

25. Secondary Outcome: Change From Baseline At Week 24 In The UFS-QoL Revised Activities Scale Score
Description: Transformed score ranges from 0 to 100 based on Likert scale (none of time, a little of time, some of the time, most of the time and all of the time). Higher scores are indicative of better health-related quality of life (high score = good). LS means and p-value for test of difference was relugolix plus E2/NETA minus placebo based on mixed-effect model with treatment, visit, region, Baseline MBL and treatment by visit interaction included as fixed effects.
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms are presented.
Time Frame: Baseline, Week 24
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 96 | 95
units on a scale | 44.4 (2.90) | 16.5 (2.94)
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 24, analysis 1]

26. Secondary Outcome: Change From Baseline In UFS-QoL Score by Health-Related Quality of Life Total Score
Description: The UFS-QoL total score was the sum of 6 subscales (concern, activities, energy/mood, control, self-conscious, and sexual function). The raw scores were transformed to normalized scores. Transformed score ranges from 0 to 100. Higher scores are indicative of better health-related quality of life (high = good).
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms are presented.
Time Frame: Baseline, Week 24
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 96 | 95
units on a scale | 37.8 (2.49) | 13.8 (2.51)
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 24, analysis 1]

27. Secondary Outcome: Number Of Responders With At Least 20 Points Increase From Baseline At Week 24 In UFS-QoL Revised Activities Scale Score
Description: as for outcome 20
Time Frame: From Baseline through Week 24
Population: All participants who were randomized to treatment and who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 125 | 129
Participants | 78 | 42
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was based on Cochran-Mantel-Haenszel test stratified by Baseline MBL volume (< 225 mL, ≥ 225 mL) and geographic region (North America, Rest of World)

28. Secondary Outcome: Change From Baseline in UFS-QoL Bleeding and Pelvic Discomfort Scale Score
Description: The Bleeding and Pelvic Discomfort Scale consists of 3 items proximal to uterine fibroids that are experienced by most participants (heavy bleeding during the menstrual period [Question 1], passing blood clots during the menstrual period [Question 2], and feeling tightness or pressure in the pelvic area [Question 5]).Transformed score ranges from 0 to 100 based on Likert scale (None of time, a little of time, some of the time, most of the time and all of the time). Lower score indicates minimal symptom severity and higher score indicates maximum symptom severity. A negative change from baseline indicates improvement.
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms are presented.
Time Frame: Baseline, Week 24
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 96 | 95
score on a scale | -51.7 (2.91) | -18.3 (2.95)
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 23, analysis 1]

29. Secondary Outcome: Number Of Responders With At Least 20 Points Decrease in UFS-QoL Bleeding And Pelvic Discomfort Scale Score
Description: Responder was defined as meeting a meaningful change threshold, set as a 20-point change from Baseline, in the Bleeding And Pelvic Discomfort Scale at Week 24 on the transformed score.
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms are presented.
Time Frame: Baseline, Week 24
Population: All participants who were randomized to treatment and who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 125 | 129
Participants | 79 | 37
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 27, analysis 1]

30. Secondary Outcome: Change From Baseline At Week 24 In The Interference Of Uterine Fibroids With Physical Activities Based On UFS-QoL Question 11
Description: Transformed score ranges from 0 to 100 based on Likert scale (None of time, a little of time, some of the time, most of the time and all of the time). Lower score indicates minimal symptom severity and higher score indicates maximum symptom severity. A negative change from baseline indicates improvement.
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms are presented.
Time Frame: Baseline, Week 24
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 96 | 95
score on a scale | -2.0 (0.14) | -0.7 (0.14)
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 24, analysis 1]

31. Secondary Outcome: Change From Baseline At Week 24 In The Interference Of Uterine Fibroids With Social Activities Based On UFS-QoL Question 20
Description: as for outcome 30
Time Frame: Baseline, Week 24
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 96 | 95
score on a scale | -1.8 (0.13) | -0.6 (0.13)
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 24, analysis 1]

32. Secondary Outcome: Change From Baseline At Week 24 In Embarrassment Caused By Uterine Fibroids Based On UFS-QoL Question 29
Description: as for outcome 30
Time Frame: Baseline, Week 24
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 96 | 95
score on a scale | -1.4 (0.14) | -0.7 (0.14)

33. Secondary Outcome: Change From Baseline At Week 24 In Symptoms Assessed Using The Patient Global Assessment (PGA) Questionnaire
Description: PGAs assessed participants' limitation in activities and the severity of symptoms due to uterine fibroids over the previous 4 weeks, as perceived by the participant. The PGA for symptoms is a 1-item questionnaire designed to assess participant's impression of the severity of their symptoms related to uterine fibroids. The PGA for function and symptoms was evaluated using a 5-point response scale (no limitation at all [1], mild limitation [2], moderate limitation [3], quite a bit of limitation [4], and extreme limitation [5]).
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms are presented.
Time Frame: Baseline, Week 24
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 80 | 84
score on a scale | -2.0 (0.14) | -0.8 (0.14)
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 24, analysis 1]

34. Secondary Outcome: Change From Baseline At Week 24 In Function Assessed Using The PGA Questionnaire
Description: as for outcome 33
Time Frame: Baseline, Week 24
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 80 | 84
score on a scale | -1.7 (0.15) | -0.8 (0.15)

35. Secondary Outcome: Participants Achieving Improvement From Baseline In PGA Questionnaire For Symptoms From Baseline At Week 24
Description: The PGAs assessed participants' limitation in activities and the severity of symptoms due to uterine fibroids over the previous 4 weeks, as perceived by the participant. The PGA for function and symptoms was evaluated using a 5-point response scale (no limitation at all [1], mild limitation [2], moderate limitation [3], quite a bit of limitation [4], and extreme limitation [5]). Category improvements for symptoms are presented. A 1-category improvement would be severe at baseline to moderate.
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms are presented.
Time Frame: From Baseline through Week 24
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 80 | 84
Participants
  1 Category improvement (-1) | 7 | 21
  3 Category improvement (-3) | 22 | 8
  2 Category improvement (-2) | 29 | 18
  4 Category improvement (-4) | 10 | 2

36. Secondary Outcome: Participants Achieving Improvement From Baseline In PGA For Uterine Fibroid-related Function From Baseline At Week 24
Description: as for outcome 35
Time Frame: From Baseline through Week 24
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 80 | 84
Participants
  1 Category improvement (-1) | 13 | 19
  2 Category improvement (-2) | 30 | 13
  3 Category improvement (-3) | 18 | 10
  4 Category improvement (-4) | 4 | 2

37. Secondary Outcome: Change From Baseline At Week 24 In The Menorrhagia Impact Questionnaire Score For Physical Activities
Description: The Menorrhagia Impact was evaluated using a 5-point response scale to assess level of improvement from Baseline to Week 24. Response scale: Not at all, 2. Slightly, 3.Moderately, 4. Quite a bit and 5. Extremely.
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms are presented.
Time Frame: Baseline, Week 24
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 94 | 95
score on a scale | -1.8 (0.14) | -0.9 (0.14)

38. Secondary Outcome: Change From Baseline At Week 24 In The Menorrhagia Impact Questionnaire Score For Social Activities
Description: as for outcome 37
Time Frame: Baseline, Week 24
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 94 | 95
score on a scale | -1.8 (0.14) | -1.0 (0.14)

39. Secondary Outcome: Number Of Participants Who Achieved A Maximum NRS Score ≤ 1 For Uterine Fibroid-associated Pain Over The Last 35 Days Of Treatment Who Had Maximum Pain Scores ≥ 4 During The 35 Days Prior To Randomization
Description: Uterine fibroid-associated pain was assessed by a pain NRS. The pain NRS is a validated, single-item, self-reported measure, which asks respondents to rank their pain on an 11-point scale as follows: 0 (no pain), 1 to 3 (mild pain), 4 to 6 (moderate pain), and 7 to 10 (severe pain).
  As per the objective of the study, the pre-specified secondary efficacy analyses compared relugolix plus E2/NETA with placebo. Therefore, only relugolix plus E2/NETA and placebo arms are presented.
Time Frame: From Baseline up to the last 35 days of treatment (up to 24 weeks)
Population: All participants who were randomized to treatment and who received at least 1 dose of study drug who had a maximum NRS score ≥ 4 at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 93 | 95
Participants | 34 | 17

40. Secondary Outcome: Number Of Participants With A ≥ 30% Reduction in NRS Score From Baseline to Last 35 Days of Treatment Who Had Maximum Pain Scores ≥ 4 At Baseline
Description: as for outcome 39
Time Frame: Baseline, Week 24
Population: All participants who were randomized to treatment and who received at least 1 dose of study drug who had a maximum NRS score ≥ 4 at baseline and had at least 28 days (80% of the last 35 days of treatment) of pain scores recorded in the e-Diary.
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 68 | 82
Participants | 48 | 34
Statistical Analysis 1: Comparison: Relugolix Plus E2/NETA (Group A) vs Placebo (Group C); Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel — [p-value comment as in outcome 27, analysis 1]

41. Secondary Outcome: Change From Baseline In Luteinizing Serum Concentration At Week 24
Description: as for outcome 20
Time Frame: Baseline, Week 24
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 92 | 93
IU/L | -3.10 (4.807) | 3.04 (13.162)

42. Secondary Outcome: Change From Baseline In Follicle Stimulating Serum Concentration At Week 24
Description: as for outcome 20
Time Frame: Baseline, Week 24
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 92 | 93
IU/L | -5.47 (9.049) | -0.67 (7.422)

43. Secondary Outcome: Change From Baseline In E2 Serum Concentration At Week 24
Description: as for outcome 20
Time Frame: Baseline, Week 24
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 93 | 90
pg/mL | -22.30 (66.552) | 39.85 (99.578)

44. Secondary Outcome: Change From Baseline In Progesterone Serum Concentration At Week 24
Description: as for outcome 20
Time Frame: Baseline, Week 24
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Relugolix Plus E2/NETA (Group A) | Placebo (Group C)
Number analyzed (Participants) | 92 | 93
ng/mL | 0.12 (3.963) | 3.48 (5.415)

ADVERSE EVENTS:
Time Frame: From Day 1 to End of Study (24 Weeks)
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/126 | 0/129
Serious Adverse Events (participants affected / at risk) | 1/126 | 2/126 | 4/129
Other Adverse Events (participants affected / at risk) | 31/126 | 67/126 | 42/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relugolix Plus E2/NETA (Group A) (N=126) | Relugolix Plus Delayed E2/NETA (Group B) (N=126) | Placebo (Group C) (N=129)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relugolix Plus E2/NETA (Group A) (N=126) | Relugolix Plus Delayed E2/NETA (Group B) (N=126) | Placebo (Group C) (N=129)
Hot flush (Vascular disorders) | 7 (7) | 44 (46) | 5 (5)
Hypertension (Vascular disorders) | 5 (5) | 7 (7) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 7 (7)
Headache (Nervous system disorders) | 11 (15) | 28 (34) | 15 (21)
Fatigue (General disorders) | 1 (1) | 7 (7) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (6) | 4 (4) | 10 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 8 (11) | 4 (6)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 3 (3) | 7 (7)

LIMITATIONS AND CAVEATS:
None reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-09-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT03103087/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT03103087/SAP_001.pdf